CLINICAL TRIAL: NCT06017726
Title: Insulin Resistance in Non-diabetic Multiple Sclerosis Patients: Prevalence, Pre and Post-treatment Effect on Clinical, Cognitive Profile, Laboratory, and Radiological Markers
Brief Title: Insulin Resistance in Egyptian Patients With Multiple Sclerosis
Acronym: IR-MS
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, doaa mokhtar mahmoud, lecturer, Assiut University
Other Study IDs: IR in Egyptian MS patients
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis; Insulin Resistance
MeSH Terms: conditions — Multiple Sclerosis; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Multiple sclerosis patients without insulin resistance: Cognitive status will be evaluated with BICAMS test. Physical disability will be evaluated by the EDSS score, 9-hole pig and 25-foot-walk test. Patients will be assessed for other comorbid conditions like fatigue and depression. Serum light chain neurofilaments as a laboratory marker for axonal degeneration will be used. brain imaging will be done with with Diffusion tensor imaging.
- Multiple sclerosis patients with treated insulin resistance: before and after treatment of insulin resistance Cognitive status will be evaluated with BICAMS test. Physical disability will be evaluated by the EDSS score, 9-hole pig and 25-foot-walk test. Patients will be assessed for other comorbid conditions like fatigue and depression. Serum light chain neurofilaments as a laboratory marker for axonal degeneration will be used. brain imaging will be done with with Diffusion tensor imaging.
  Interventions: Other: treatment of insulin resistance with appropriate modality according to each patient
- Multiple sclerosis patients with untreated insulin resistance: at the end of the 1st and 2nd year of the study, Cognitive status will be evaluated with BICAMS test. Physical disability will be evaluated by the EDSS score, 9-hole pig and 25-foot-walk test. Patients will be assessed for other comorbid conditions like fatigue and depression. Serum light chain neurofilaments as a laboratory marker for axonal degeneration will be used. brain imaging will be done with with Diffusion tensor imaging.

INTERVENTIONS:
Other: treatment of insulin resistance with appropriate modality according to each patient — insulin resistance will be treated with either diet alone or combined diet and appropriate pharmacological treatment with the net result of normalization of HOMA IR index
  Groups: Multiple sclerosis patients with treated insulin resistance

SUMMARY:
The goal of this three-phase interventional study is to determine the prevalence of Insulin resistance in non-diabetic patients with multiple sclerosis in Egypt

The main questions it aims to answer are:

1. what is the prevalence of insult resistance among Egyptian patients with Multiple sclerosis?
2. what are the effects of insulin resistance on multiple sclerosis disease activity and progression
3. what are the effects of treating insulin resistance on multiple sclerosis disease activity and progression participants with MS will be tested for IR to determine its prevalence, in the 2nd phase a group of MS patients with IR will be compared with another control group of MS patients without IR for clinical, laboratory, and radiological markers of disease activity and progression twice at baseline and after 1 year. in the 3rd phase, patients with IR will be divided into 2 groups one who will receive appropriate treatment for IR and the other group without treatment of IR and will be compared by the end of the 2nd year for clinical, laboratory and radiological markers of disease activity and progression

DETAILED DESCRIPTION:
In this longitudinal, three-phase, case-control, interventional study, with 250 patients with multiple sclerosis diagnosed according to the 2017 McDonald's criteria will be enrolled. Frist diagnosis of cases of insulin resistant MS patient out of the total sample of MS through estimation of fasting blood glucose, insulin level, and homeostatic model assessment of insulin resistance (HOMA-IR) index. Other supportive indices like waste circumference, hemoglobin A1c, and lipid profile will be used. At the end of first phase, prevalence of IR and associated metabolic syndrome will be determined. In the second phase of the study, patients will be divided into two groups with and without IR. Cognitive status will be evaluated with BICAMS test. Physical disability will be evaluated by the EDSS score, 9-hole pig and 25-foot-walk test. Patients will be assessed for other comorbid conditions like fatigue and depression. Serum light chain neurofilaments as a laboratory marker for axonal degeneration will be used. Diffusion tensor imaging with a fully automated too (volbrain) will be used. Patients in the second phase of the study will be evaluated both at baseline and after one year. In the third phase, patients with IR will be divided randomly into two equal groups (1:1) using closed envelope: intervention group who will receive appropriate treatment for IR and a control group with placebo treatment (without IR treatment) and by the end of the second year all groups will be evaluated blindly using the same evaluating measures (clinical, laboratory and radiological)

ELIGIBILITY:
Inclusion Criteria:

* seventy patients aged 18-50 years old of both sex fulfilling the revised McDonald's Criteria for diagnosis of multiple sclerosis 2017 of different phenotypes (relapsing-remitting, primary progressive, and secondary progressive), will be recruited during their follow-up visits to our MS unit.

Exclusion Criteria:

* • Recent MS relapse or use of corticosteroids in the past 3 months

  * patients with a systemic disease like diabetes mellitus, hypertension, cardiac disease, liver or renal disease or alcoholic patients
  * patients who are on a specific diet.
  * patients using any anti-inflammatory drugs, cholesterol-lowering agents, estrogen replacement therapy, steroid therapy or other drugs that could affect the metabolic profile.
  * Patients with non-MS demyelinating disorders like NMOSD and MOGAD.
  * Patients who failed to commit to regular follow-ups.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: multiple sclerosis patients diagnosed according to the revised McDonald's Criteria for diagnosis of multiple sclerosis 2017 of different phenotypes (relapsing-remitting, primary progressive, and secondary progressive)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
prevalence of insulin resistance among Egyptians with multiple sclerosis | this will be determined in the first 2 months of the study (phase 1 of the study)
  to determine the prevalence of Insulin resistance among Egyptian patients with multiple sclerosis using the homeostatic model assessment of insulin resistance (HOMA-IR) index

SECONDARY OUTCOMES:
effect of insulin resistance on Multiple sclerosis disease activity | this evaluation will be done at 2 points; at the beginning and the end of the first year of the study (phase 2)
  disease activity (indicated by either annualized relapse rate or radiological activity) will be compared between MS patients with and without Insulin resistance
effect of insulin resistance on Multiple sclerosis disease progression | this evaluation will be done at 2 points; at the beginning and the end of the first year of the study (phase 2)
  disease progression (indicated by either changes in BICAMS scores, or radiological markers of progression) will be compared between MS patients with and without Insulin resistance
effect of treating insulin resistance on Multiple sclerosis disease activity | this evaluation will be done at 2 points; at the beginning and the end of the second year of the study (phase 3)
  disease activity (indicated by either annualized relapse rate or radiological activity) will be compared between MS patients with treated and untreated Insulin resistance
effect of treating insulin resistance on Multiple sclerosis disease progression | this evaluation will be done at 2 points; at the beginning and the end of the second year of the study (phase 3)
  disease progression (indicated by either changes in BICAMS scores or radiological markers of progression) will be compared between MS patients with treated and untreated Insulin resistance

IPD SHARING:
Plan to Share IPD: No